CLINICAL TRIAL: NCT02328625
Title: Scleroderma Treatment With Celution Processed Adipose Derived Regenerative Cells (ADRCs) Registry
Brief Title: Scleroderma Treatment With Celution Processed ADRCs Registry
Acronym: STAR
Status: Withdrawn | Type: Observational
Why Stopped: Corporate decision
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: STAR Registry
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Scleroderma
Keywords: Scleroderma; Device; ADRCs; adipose derived regenerative cells; hand
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry study will assess the safety and performance of the Celution Device in the processing of an autologous graft consisting of adipose derived regenerative cells (ADRCs) in the treatment of hand scleroderma.

DETAILED DESCRIPTION:
This registry study will assess the safety and performance of the Celution System in preparation of adipose derived regenerative cells in the treatment of scleroderma affecting the hands. This will be a multi-center, multi-national study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of scleroderma and presence of hand scleroderma
* Cochin score ≥ 20 units

Exclusion Criteria:

* Body Mass Index < 17 kg/m2
* Infection in any finger
* Stable medications for the treatment of scleroderma for ≥ 1 month
* Pregnant or lactating status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive or have received ADRCs prepared by Celution to treat hand scleroderma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in Cochin score | Day 90

SECONDARY OUTCOMES:
Change in Cochin score | Days 30 and 180
Scleroderma Health Assessment Questionnaire (SHAQ) | Days 7, 30, 90 and 180
Physician and Patient Global Assessment | Days 7, 30, 90 and 180
Raynaud's Condition Score | Days 7, 30, 90 and 180
EQ-5D | Days 7, 30, 90 and 180

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, Study Chair — Cytori Therapeutics